CLINICAL TRIAL: NCT02598765
Title: Micro vs. Standard Trabeculectomy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: Seva Foundation (Other); Lumbini Eye Institute and Research Centre (Other)
Responsible Party: Principal Investigator, Jeremy Keenan, Associate Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-16075
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Glaucoma
Keywords: Glaucoma; Trabeculectomy; Eye Disease; Intraocular Pressure; Visual Acuity
MeSH Terms: conditions — Glaucoma; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Trabeculectomy (Active Comparator): Patients in the Standard Trabeculectomy arm will undergo regular trabeculectomy
  Interventions: Procedure: Standard Trabeculectomy
- Microtrabeculectomy (Experimental): Patients in the Microtrabeculectomy arm will undergo microtrabeculectomy
  Interventions: Procedure: Microtrabeculectomy

INTERVENTIONS:
Procedure: Standard Trabeculectomy — Fornix-based trabeculectomy with a 3x4 mm scleral flap.
  Arms: Standard Trabeculectomy
Procedure: Microtrabeculectomy — Fornix-based trabeculectomy with a 2x2 mm scleral flap.
  Arms: Microtrabeculectomy

SUMMARY:
The purpose of this study is to determine the reduction in intraocular pressure and cumulative incidence of complications between the standard and micro trabeculectomy surgeries 3 months after surgery.

DETAILED DESCRIPTION:
This study is a randomized, double-masked (study participants and outcome assessors) trial. During the enrollment period, consecutive patients from LEI who are planning to have trabeculectomy surgery and who meet the study enrollment criteria will be randomized to receive standard trabeculectomy or microtrabeculectomy. The primary outcome is complications and change in intraocular pressure after a 3 month follow-up period. We will perform subgroup analyses by stratifying the population according to skin pigmentation to determine whether pigmentation is a predictor of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 40
* Planning to have a trabeculectomy

Exclusion Criteria:

* Life threatening or debilitating disease
* Inability to complete necessary exams and/or ocular disease that would preclude assessment of intraocular pressure, visual field, or optic disc
* Contralateral eye already enrolled in study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of complications | 3 months after surgery
  Comparison of the cumulative incidence of complications between the treatment groups (regular and micro trabeculectomy) 3 months after surgery

SECONDARY OUTCOMES:
Reduction in intraocular pressure | 3 months after surgery
  Comparison of the reduction in intraocular pressure between the treatment groups (regular and micro trabeculectomy) 3 months after surgery
Cumulative incidence of complications | 6 and 12 months after surgery
  Cumulative incidence of complications 6 months and 12 months after surgery will be compared between the treatment groups
Reduction of intraocular pressure | 6 and 12 months after surgery
  Reduction of intraocular pressure 6 months and 12 months after surgery will be compared between the treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy D Keenan, MD, MPH, Principal Investigator — F. I. Proctor Foundation, UCSF
Locations (1):
- Lumbini Eye Institute, Nepal, Siddharthanagar, Nepal